CLINICAL TRIAL: NCT03925688
Title: Assessment of Heterotopic Ossification of Elbow Joint in Relation of Serum Uric Acid: a Retrospective Study.
Brief Title: Assessment of Heterotopic Ossification of Elbow Joint in Relation of Serum Uric Acid.
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: I2019001071
Record Dates: First submitted 2019-04-21; First posted 2019-04-24 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Heterotopic Ossification
Keywords: heterotopic ossification; serum uric acid，; elbow joint
MeSH Terms: conditions — Ossification, Heterotopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- without heterotopic ossification: There had not existed radiographic evidences of heterotopic ossification.
- with heterotopic ossification: There had existed radiographic evidences of heterotopic ossification or formatted ectopic lamellar bone.

SUMMARY:
Heterotopic ossification (HO) is a common complication after surgical repair of elbow trauma. Uric acid is the end-product of purine metabolism that has any physiological and pathogenic potential functions. However, the relationship of HO and uric acid has not been explored up to now. This study aimed to assess the relationship of HO and uric acid. The investigators retrospectively reviewed the demographics of participants who undergone the surgery for elbow trauma in our hospital between January 2012 and December 2018. One hundred participants included in our study. The participants were divided into two groups by the existing HO or not. The serum uric acid between both groups were compared by using the independent samples student T tests.

DETAILED DESCRIPTION:
The investigators retrospectively analyzed the demographics of these participants in our hospital who underwent the surgery after trauma of elbow joint between January 2012 and December 2018. All of the participants had a previous history of elbow joint fractures including distal humerus fracture or proximal ulna fracture or capitulum radii fracture or elbow fracture dislocation. According to X ray or CT scan, the participants were divided into two groups. One group the participants had not existed radiographic evidence of heterotopic ossification or formatted ectopic lamellar bone. And the other group is the participants with radiographic evidence of heterotopic ossification. And we recorded patient serum uric acid, sex and age, Body Mass Index (BMI), the situation of joint trauma and comorbid conditions including diabetes mellitus or impaired blood glucose, gout, metabolic syndrome, osteoporosis and various vitamin deficiency diseases. Moreover, the grades of heterotopic ossification were recorded for all patients according to Hastings and Graham Classification System for Heterotopic Ossification at the Elbow Joint.

ELIGIBILITY:
Inclusion Criteria:

* Have a previous history of elbow joint fracture or dislocation that conform to its manifestations and signs. And it is diagnosed by X-ray test. HO must accord with the relative diagnostic criteria5 and have imaging evidences of heterotopic ossification.
* Have complete clinical and imaging dates.
* The age>18 and no gender limitation.
* The patient is being a relatively stable physical and mental state without acute injection or diseases.

Exclusion Criteria:

* Have a history of diabetes mellitus or impaired blood glucose, metabolic syndrome and gout or renal dysfunction (creatinine ≥ 1.5 mg/dL) that apparently influence glucose, lipid and protein metabolic of the body.
* Have a history of taking drugs that can influence uric acid metabolic including gout suppressant, diuretic, small-dose aspirin (75~300mg/d) or large-dose aspirin (>3g/d), anti-tuberculosis drugs, immunosuppressor, nicotinic acid and anti-tumor drugs such as cyclophosphamide and so on.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population came from The Second Affiliated Hospital of Zhejiang University.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
serum uric acid value | the outcome of serum uric acid can acquire within half a day.
  The serum uric acid was measured by standard equipment in the laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Jian'an Wang, Ph.D, Study Chair — Zhejiang University
Locations (1):
- Institutional Review Board of The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China